CLINICAL TRIAL: NCT00665470
Title: Phase II Study in Patients With Metastatic Melanoma Using a Non-Myeloablative Lymphocyte Depleting Regimen of Chemotherapy Followed by Infusion of gp100 Reactive Peripheral Blood Lymphocytes (PBL) and High or Low Dose Aldesleukin
Brief Title: Chemotherapy Followed by gp100 Lymphocytes and Aldesleukin to Treat Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Udai Kammula, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080104; 08-C-0104
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Results first posted 2013-01-22 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Skin Cancer; Metastatic Melanoma
Keywords: Malignant Melanoma; HLA-A2; Immunotherapy; Clinical Response; Skin Cancer
MeSH Terms: conditions — Skin Neoplasms; Melanoma | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort I - high dose Aldesleukin (Experimental): Patients receive high-dose aldesleukin intravenous (IV) over 15 minutes every 8 hours beginning within 24 hours after peripheral blood lymphocyte (PBL) infusion and continuing for up to 5 days (maximum of 15 doses).
  Interventions: Drug: Aldesleukin
- Cohort II - low dose Aldesleukin (Experimental): Beginning within 24 hours after peripheral blood lymphocyte (PBL) infusion, patients receive low-dose aldesleukin subcutaneous (SC) once daily 5 days a week for up to 6 weeks.
  Interventions: Drug: Aldesleukin

INTERVENTIONS:
Drug: Aldesleukin — High-dose aldesleukin intravenous (IV) over 15 minutes every 8 hours beginning within 24 hours after peripheral blood lymphocyte (PBL) infusion and continuing for up to 5 days (maximum of 15 doses).
  Receive low-dose aldesleukin subcutaneously (SC) once daily 5 days a week for up to 6 weeks

SUMMARY:
Background:

This study uses a new experimental procedure for treating melanoma that uses the patient's own lymphocytes (type of white blood cell), which are specially selected to target and destroy their tumor.

Objectives:

To determine whether this experimental treatment can cause the patient's tumor to shrink.

To test the safety of the treatment and its effects on the immune system.

Eligibility:

Patients with metastatic melanoma 18 years of age and older for whom standard treatments are not effective or who cannot take high-dose interleukin-2 (IL-2).

Patients must have the tissue type human leukocyte antigens (HLA-A)0201.

Design:

Workup: Patients have scans, x-rays, laboratory tests, and other tests as needed.

Patients have leukapheresis (a procedure for collecting lymphocytes that is similar to collecting whole blood) to collect cells for laboratory treatment and later reinfusion.

Chemotherapy: Patients have low-dose chemotherapy for 1 week to prepare the immune system to receive the cultured lymphocytes.

Cell infusion and IL-2 treatment: Patients receive the lymphocytes by infusion through a vein and then either high-dose IL-2 infused through a vein or low-dose IL-2 injected under the skin. High-dose IL-2 is given as infusions through a vein every 8 hours for up to 15 doses. Low-dose IL-2 is given as injections under the skin daily for 5 days, followed by a 2-day rest, with this regimen repeated for a total of 5 weeks.

Recovery: Patients rest for 1 to 2 weeks to recover from the effects of chemotherapy and IL-2.

Tumor biopsy: Patients may be asked to have a biopsy (removal of a small piece of tumor) after receiving treatment to look at the effects of treatment in the tumor.

Follow-up: After treatment is completed, patients return to the clinic for physical examinations, review of side effects, laboratory tests and scans every 1 to 6 months until the disease worsens.

Retreatment: Patients whose tumor did not grow after treatment or showed evidence of shrinking may be able to be retreated if their tumor begins to grow. They receive the same regimen of chemotherapy, lymphocyte infusion and IL-2 treatment....

DETAILED DESCRIPTION:
Background:

* Tumor infiltrating lymphocytes (TIL) transfer studies in patients with metastatic melanoma following lymphodepletion have resulted in 50% objective response rates with a 10-15% rate of complete responses.
* Pre-clinical and clinical studies of adoptive immunotherapy have suggested that effective lymphocytes for transfer have high avidity for the target antigen, undergo limited in vitro antigen and IL-2 stimulation, and have high expression of cluster of differentiation 27+ (CD27+).
* We have developed a novel in vitro strategy using high throughput polymerase chain reaction (PCR) screening to rapidly isolate low frequency antigen specific cluster of differentiation 8+ (CD8+) T cells from the peripheral blood repertoire that have these characteristics, and that recognize the gp100:154-162 epitope, an abundantly expressed melanoma antigen, presented by human leukocyte antigens (HLAA2) on the tumor surface.
* The current proposed transfer of gp100:154-162 reactive lymphocytes administered in conjunction with a lymphodepleting preparative regimen and aldesleukin would represent a significantly novel approach to adoptive immunotherapy.

Objectives:

* To determine whether gp100:154-162 reactive cluster of differentiation 4+ (CD4+) T cell depleted lymphocytes infused in conjunction with the administration of high-dose aldesleukin or low-dose aldesleukin may result in clinical tumor regression in patients with metastatic melanoma receiving a non-myeloablative lymphoid depleting preparative regimen.
* To evaluate the safety of the treatment in patients receiving the non-myeloablative conditioning regimen, cell transfer, and high-dose or low-dose aldesleukin.
* To determine the survival in patients, of infused cells following the administration of the non-myeloablative regimen, using analysis of the sequence of the variable region of the T cell receptor or flow cytometry (fluorescence activated cell sorting-FACS).

Eligibility:

-Patients with refractory metastatic melanoma who are greater than or equal to 18 years of age, are HLA-A2+, who have gp100:154-162 reactive peripheral blood lymphocytes available and are physically able to tolerate non-myeloablative chemotherapy. Patients must be refractory to prior high dose aldesleukin treatment if they are medically eligible to receive it. Patients who can tolerate high-dose aldesleukin will receive it with cell infusion; those who cannot tolerate high-dose will receive low-dose aldesleukin.

Design:

* Patients will receive a non-myeloablative lymphocyte depleting preparative regimen consisting of cyclophosphamide (60 mg/kg/day X 2 days intravenous (IV)), fludarabine (25 mg/m^2/day IV X 5 days).
* Patients will receive intravenous adoptive transfer of gp100:154-162 reactive peripheral blood lymphocytes (minimum 1 X 10^9) and up to a maximum of 3 X 10^11) lymphocytes) followed by high-dose intravenous (IV) aldesleukin (720,000 IU/kg/dose every 8 hours for up to 15 doses) or low-dose subcutaneous (SQ) aldesleukin (125,000 IU IL-2/kg/dose for 5 days for 6 weeks with 2 days rest per week).
* A complete evaluation of evaluable lesions will be conducted 4-6 weeks after the last dose of aldesleukin in the high dose arm and 2-4 weeks after the last dose of aldesleukin in the low dose arm. Patients will be enrolled into two cohorts. The cohort receiving high dose aldesleukin will be conducted using a small optimal two-stage Phase II design, initially 21 patients will be enrolled, and if two or more of the first 21 patients has a clinical response (partial response (PR) or complete response (CR)), accrual will continue to 41 patients, targeting a 20% goal for objective response. For the cohort who will receive low dose aldesleukin, the study will be conducted as a Minimax two-stage phase II trial. Initially 12 evaluable patients will be enrolled to this cohort, and if 1 or more the first 12 have a response, then accrual would continue until a total of 21 patients, targeting a 20% goal for objective response.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable metastatic melanoma. The diagnosis of metastatic melanoma and positivity for gp100 will be confirmed by the Laboratory of Pathology of the the National Cancer Institute (NCI).
2. Patients must be refractory to high dose aldesleukin treatment if they are medically eligible to receive it. Patients with noncutaneous melanoma are not required to be refractory to high dose aldesleukin.
3. gp100:154-162 reactive peripheral blood lymphocytes derived from a

   leukapheresis.
4. HLA-A*0201 positive.
5. Greater than or equal to 18 years of age.
6. Willing to practice birth control during treatment and for four months after receiving the preparative regimen.
7. Life expectancy of greater than three months.
8. Willing to sign a durable power of attorney.
9. Able to understand and sign the Informed Consent Document.
10. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1 for the high dose aldesleukin cohort or ECOG 0, 1 or 2 for the low dose aldesleukin cohort.
11. Hematology:

    * Absolute neutrophil count greater than 1000/mm^3 without support of filgrastim
    * Normal white blood cell (WBC) (greater than 3000/mm^3).
    * Hemoglobin greater than 8.0 g/dl
    * Platelet count greater than 100,000/mm^3.
12. Serology:

    * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B or hepatitis C.
13. Chemistry:

    * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than less or equal to 2.5 times the upper limit of normal.
    * Serum creatinine less than or equal to 1.6 mg/dl.
    * Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3 mg/dl.
14. Negative pregnancy test in women of child bearing potential because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
15. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo). Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria in Section 2.1.1.
16. Six weeks must have elapsed since prior cytotoxic T-lymphocyte antigen 4 (anti-CTLA4) antibody therapy to allow antibody levels to decline.
17. Patients who have previously received anti-CTLA4 antibody and experienced treatment must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
2. Systemic steroid therapy required.
3. For patients receiving high dose IL-2 only: Active systemic infections, coagulation disorders or other active major medical illnesses of the cardiovascular, respiratory or immune system, as evidenced by a positive stress thallium or comparable test, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
4. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
5. Opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. The following patients will be excluded from the high-dose IL-2 arm (but will be eligible for the low-dose arm):

   1. History of coronary revascularization or ischemic symptoms
   2. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45%.
   3. Documented LVEF of less than or equal to 45% tested in patients with:

      * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
      * Age greater than or equal to 60 years old
   4. Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

      * A prolonged history of cigarette smoking (20 pk/yrs of smoking)
      * Symptoms of respiratory dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joohee Sul, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Atkins MB, Kunkel L, Sznol M, Rosenberg SA. High-dose recombinant interleukin-2 therapy in patients with metastatic melanoma: long-term survival update. Cancer J Sci Am. 2000 Feb;6 Suppl 1:S11-4. PMID 10685652
- [Background] Gogas HJ, Kirkwood JM, Sondak VK. Chemotherapy for metastatic melanoma: time for a change? Cancer. 2007 Feb 1;109(3):455-64. doi: 10.1002/cncr.22427. PMID 17200963
- [Background] Rosenberg SA. Progress in human tumour immunology and immunotherapy. Nature. 2001 May 17;411(6835):380-4. doi: 10.1038/35077246. PMID 11357146
- [Derived] Wang A, Chandran S, Shah SA, Chiu Y, Paria BC, Aghamolla T, Alvarez-Downing MM, Lee CC, Singh S, Li T, Dudley ME, Restifo NP, Rosenberg SA, Kammula US. The stoichiometric production of IL-2 and IFN-gamma mRNA defines memory T cells that can self-renew after adoptive transfer in humans. Sci Transl Med. 2012 Aug 29;4(149):149ra120. doi: 10.1126/scitranslmed.3004306. PMID 22932225

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All patients were enrolled into cohort I because all patients were able to receive high dose IL-2.
Period: Overall Study
Arm/Group | Cohort I - High Dose Aldesleukin | Cohort II - Low Dose Aldesleukin
Started | 10 | 0
Completed | 10 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I - High Dose Aldesleukin | Cohort II - Low Dose Aldesleukin | Total
Number analyzed (Participants) | 10 | 0 | 10
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 9 |  | 9
  >=65 years | 1 |  | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.36 (9.23) |  | 54.36 (9.23)
Gender [Number; unit: participants]
  Female | 2 |  | 2
  Male | 8 |  | 8
Ethnicity (NIH/OMB) [Number; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 10 |  | 10
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Number; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 9 |  | 9
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Response is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is a disappearance of all target lesions. Partial response (PR) is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progression (PD) is at least a 20% increase in the sum of LD of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more lesions. Stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD.
Time Frame: 30 months
Measure: Number; unit: Participants
Arm/Group | Cohort I - High Dose Aldesleukin | Cohort II - Low Dose Aldesleukin
Number analyzed (Participants) | 10 | 0
Participants
  Complete Response | 0 |
  Partial Response | 0 |
  Progression | 8 |
  Stable Disease | 2 |

2. Primary Outcome: Toxicity as Assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) V3.0
Description: Here is the number of participants with adverse events. For a detailed list of participants with adverse events, see the adverse event module.
Time Frame: 16 months
Measure: Number; unit: Participants
Arm/Group | Cohort I - High Dose Aldesleukin | Cohort II - Low Dose Aldesleukin
Number analyzed (Participants) | 10 | 0
Participants | 10 |

ADVERSE EVENTS:
Arm/Group | Cohort I - High Dose Aldesleukin | Cohort II - Low Dose Aldesleukin
Serious Adverse Events (participants affected / at risk) | 3/10 | 0/0
Other Adverse Events (participants affected / at risk) | 10/10 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I - High Dose Aldesleukin (N=10) | Cohort II - Low Dose Aldesleukin (N=0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (General disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I - High Dose Aldesleukin (N=10) | Cohort II - Low Dose Aldesleukin (N=0)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (5) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Nervous system disorders) | 2 (2) | 0 (0)
Creatinine increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 5 (5) | 0 (0)
Febrile neutropenia (Infections and infestations) | 5 (6) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, infection: klebsiella pneumoniae (Infections and infestations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 10 (12) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 10 (11) | 0 (0)
Platelet count decreased (Blood and lymphatic system disorders) | 10 (11) | 0 (0)
Rash maculo-papular (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
White blood cell decreased (Blood and lymphatic system disorders) | 10 (11) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No